CLINICAL TRIAL: NCT06898086
Title: Treatment of Severe Aortic Stenosis With Transfemoral TAVI With or Without Coronary Angiogram During Diagnostic Work-up (PURE TAVI)
Brief Title: Transfemoral TAVI With or Without Coronary Angiogram in Patients With Severe Aortic Stenosis (PURE TAVI)
Acronym: PURETAVI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rede Optimus Hospitalar SA (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RO-240905
Record Dates: First submitted 2025-03-20; First posted 2025-03-27 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Severe Aortic Stenosis
Keywords: PURE TAVI
MeSH Terms: conditions — Aortic Valve Stenosis | interventions — Transcatheter Aortic Valve Replacement

STUDY DESIGN:
Intervention Model Description: Participants are randomly assigned in a 1:1 ratio to a TAVI pathway with routine coronary angiography with or without revascularization is included or to a pathway without routine coronary angiography, and both groups are followed in parallel.
Masking Description: This is an open-label trial. Neither participants nor clinicians are masked to the treatment allocation because the performance of coronary angiography cannot be blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): (omission of coronary angiography prior to or during TAVI, unless suspicion of potentially revascularization-indicating stenosis of the left main stem based on the TAVI-CT);
  Interventions: Device: Transcatheter aortic valve implantation
- Control group (Active Comparator): (coronary angiography with or without PCI prior to TAVI).
  Interventions: Device: Transcatheter aortic valve implantation

INTERVENTIONS:
Device: Transcatheter aortic valve implantation — Transcatheter aortic valve implantation using the CE-certified Myval™ transcatheter heart valve series

SUMMARY:
This study will be conducted in patients with severe aortic stenosis who are referred for transcatheter aortic valve implantation (TAVI). TAVI is the recommended treatment for severe aortic stenosis. Currently, before undergoing TAVI, most patients undergo a coronary angiography to check whether the coronary arteries are blocked and to assist in appropriate valve sizing. If significant blockages are detected, they are treated before or during TAVI.

However, many patients who undergo TAVI are older and often have additional cardiovascular conditions such as hypertension, diabetes, or obesity. These comorbidities increase the risk of complications related to coronary angiography, including kidney injury from contrast dye, bleeding, and vascular complications at the access site. As such, it remains uncertain whether routine coronary angiography is necessary for all patients undergoing TAVI, particularly those without symptoms suggestive of myocardial ischemia.

This study aims to determine whether a TAVI treatment pathway without prior coronary angiography is non-inferior to the standard pathway that includes routine coronary angiography, with or without revascularization, in patients with severe aortic stenosis who do not have typical angina symptoms (defined as Canadian Cardiovascular Society Class <3). "Non-inferior" means the study seeks to show that omitting routine coronary angiography is at least as effective and safe as the standard approach.

All participants will receive a CE-certified Myval™ balloon-expandable transcatheter heart valve. This device is commercially available and designed to provide accurate positioning and reliable valve function.

This is a multicentre, investigator-initiated clinical study sponsored by Rede Optimus (RO), Alte Steinhauserstrasse 1, 6330 Cham, Switzerland. RO conducts independent research to address unresolved questions in vascular medicine. The study is financially supported by Meril Life Sciences Pvt. Ltd., Bilakhia House, Survey No.135/139, Muktanand Marg, Chala, Vapi 396191, Gujarat, India.

Approximately 620 patients will be enrolled across 20 centres in 7 European countries. The total study duration is expected to be 42 months, with an 18-month enrollment period and 24-month follow-up for each participant.

DETAILED DESCRIPTION:
Severe aortic stenosis is a progressive and potentially life-threatening condition in which the aortic valve becomes narrowed and obstructs blood flow from the heart. Transcatheter aortic valve implantation (TAVI) has become an established therapy for patients with severe symptomatic aortic stenosis who are not suitable for surgical valve replacement or are at increased surgical risk.

In contemporary practice, many patients undergo routine invasive coronary angiography prior to TAVI to evaluate for obstructive coronary artery disease and perform coronary revascularization when indicated. However, coronary angiography increases exposure to procedural risks, including bleeding, vascular complications, and contrast associated acute kidney injury. These risks are particularly relevant in the elderly population commonly undergoing TAVI, who may have multiple comorbidities. Emerging clinical evidence suggests that routine pre-procedural coronary angiography may not confer significant clinical benefit in all TAVI candidates, especially in those without clear symptoms of myocardial ischemia. In addition, modern transcatheter valve systems, including the balloon-expandable Myval device used in this study, are designed to allow coronary access after implantation if coronary intervention becomes necessary.

The PURE-TAVI study is a multicenter, prospective, randomized, controlled, investigator-initiated trial designed to evaluate whether a management pathway without routine pre-procedural coronary angiography is non-inferior to the standard pathway that includes routine coronary angiography with or without revascularization prior to TAVI. Eligible patients have severe aortic stenosis and are planned for transfemoral TAVI and do not report angina suggestive of high-risk coronary artery disease (Canadian Cardiovascular Society class less than 3). Approximately 620 patients across about 20 sites in Europe will be randomized in a 1:1 ratio to either standard care with routine coronary angiography and revascularization when needed or a selective approach avoiding coronary angiography unless strongly indicated by clinical or imaging findings.

All patients will receive the CE-marked, commercially available Myval transcatheter heart valve system. The trial is open-label. An independent clinical events committee will adjudicate key safety and efficacy endpoints.

The primary objective is to determine whether omission of routine coronary angiography prior to TAVI is non-inferior to the standard invasive diagnostic strategy in terms of major adverse clinical events at 12 months. The composite primary outcome includes all-cause mortality, myocardial infarction, stroke, acute kidney injury, heart failure hospitalization, and major vascular or major bleeding complications. Secondary objectives include assessment of individual clinical endpoints, need for unplanned coronary angiography or revascularization during follow-up, functional status, health-related quality of life, echocardiographic valve performance, and resource utilization.

Participants will be followed at hospital discharge, 6 months, 12 months, and 24 months. The total study duration is approximately 42 months, including an 18-month enrollment period and 24-month follow-up. This Investigator Initiated study is sponsored by Rede Optimus, Switzerland, with funding support from Meril Life Sciences. All procedures and data collection will be conducted in compliance with Good Clinical Practice, the Declaration of Helsinki, and applicable regulatory requirements.

This study aims to provide high-quality evidence on whether a simplified pre-TAVI diagnostic strategy avoiding routine invasive coronary angiography is safe and clinically effective. Results may support optimization of pre-TAVI assessment practices, reduce unnecessary invasive procedures and contrast exposure, and potentially streamline care pathways for patients with severe aortic stenosis undergoing TAVI.

ELIGIBILITY:
Inclusion Criteria:

* Patient is older than 18 years with severe AS considered for TAVI by a multidisciplinary heart team.
* Patient is candidate for transfemoral TAVI as per local standards and current guidelines.
* Patient is willing and capable to give written consent to participate to the trial and confirmed to be able to attend the expected follow up visits.

Exclusion Criteria:

* Patient had a coronary angiogram with or without PCI and/or coronary CT and/or CABG within last 5 years.
* Left main PCI in the medical history
* Patient has CCS of 3 or more.
* Patient has left ventricular ejection fraction <30%.
* Patients in whom TAVI through femoral access is ad priori not possible based on clinical assessment or medical history
* Patient has been treated for acute myocardial infarction within 30 days before randomization.
* Patient has a planned open-heart surgery.
* Patient has a life expectancy less than 1 year due to other severe non-cardiac disease.
* Patient is participating in another clinical study with an investigational product that has not yet completed the follow up period.
* Patient has received previous treatment for aortic valve implantation or replacement.
* Female patient who is pregnant at the time of inclusion and female patient of childbearing potential

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 620 (Estimated)
Dates: Start 2025-08-08 (Actual); Primary Completion 2027-10-30 (Estimated); Study Completion 2028-10-30 (Estimated)

PRIMARY OUTCOMES:
Composite of all-cause death, spontaneous or periprocedural myocardial infarction, etc | at 12-months follow-up
  Composite of all-cause death, spontaneous or periprocedural myocardial infarction, urgent revascularization during unplanned hospitalization, readmission for heart failure, acute renal injury, major or life-threatening or disabling bleeding, major vascular complication, or any stroke at 12-months follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Dr. William Wijns, Professor, Study Chair; Dr. Gabor G Toth, Professor, Study Chair; Dr. Felix Mahfoud, Professor, Study Chair; Flavio Ribichini, Professor, Study Chair; Dr. Emanuele Barbato, Professor, Study Chair; Dr. Peter Jüni, Professor, Study Chair
Locations (23):
- Austria (2):
  - Medical University Graz, Graz
  - Klinikum Klagenfurt am Wörthersee, Klagenfurt
- Czechia (2):
  - Královské Vinohrady University Hospital, Prague
  - Nemocnice Na Homolce, Prague
- France (2):
  - Institut Arnault Tzanck, Nice
  - Clinique Pasteur, Toulouse
- Germany (5):
  - Universitätsklinikum Düsseldorf, Düsseldorf, North Rhine-Westphalia
  - Elisabeth Krankenhaus Essen, Essen
  - Universitätsklinikum Freiburg- Universitäts-Herzzentrum Campus Bad Krozingen, Freiburg im Breisgau
  - Universitätsklinikum Schleswig-Holstein - Campus Lübeck, Lübeck
  - Universitätsklinikum Ulm, Ulm
- Italy (7):
  - IRCCS ISMETT Palermo, Palermo, Basel-Stadt
  - AOUP- Azienda Ospedaliera Universitaria Pisana, Pisa, Basel-Stadt
  - Azienda Ospedaliero Policlinico Universitaria G. Rodolico- San Marco Catania, Catania
  - Ospedale dell'Angelo - ULSS 3 Serenissima, Mestre
  - Fondazione Policlinico Universitario Campus Biomedico, Roma
  - Azienda Ospedaliera Universitaria Senese, Siena
  - Azienda Sanitaria Universitaria Integrata di Trieste, Trieste
- Netherlands (3):
  - Stichting Amsterdam UMC, Amsterdam
  - OLVG Hospital Amsterdam, Amsterdam
  - Clinical Trial Center Maastricht B.V, Maastricht
- Switzerland (2):
  - University Hospital Basel, Basel, Canton of Basel-City
  - University Hospital Zurich, Zurich

IPD SHARING:
Plan to Share IPD: Undecided